CLINICAL TRIAL: NCT02582437
Title: The Effect of Chronic Opioid Use on Minimum Alveolar Concentration of Sevoflurane for Maintaining Bispectral(BIS) Index Below 50 ; Prospective, Blind Study
Brief Title: MAC Bipsectral Index Below 50 for Chronic Opioid User
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Cancer Center, Korea (Other Government)
Responsible Party: Principal Investigator, Oh Tak Kyu, Anesthesiologist, National Cancer Center, Korea
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NCC2015-0147
Record Dates: First submitted 2015-10-16; First posted 2015-10-21 (Estimated); Last update posted 2015-10-21 (Estimated); Status verified 2015-10

CONDITIONS: Anesthesia
Keywords: Minimum Alveolar Concentration
MeSH Terms: interventions — Health Records, Personal

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chronic Opioid User (Experimental): The patients (ASA class I-III) who receive elective surgery s aging between 41 and 69 and signed in informed consent to participate in this trial voluntarily.
  The Patients who use opioid medication daily and regularly immediately before the day of surgery for more than four weeks. The minimum criteria for opioid dose in the intervention goup is oral morphine 20mg per day: Morphine Equivalent Daily Dose(MEDD)
  Interventions: Other: History for opioid use
- Opioid Naive patient (No Intervention): The patients (ASA class I-III) who receive elective surgery aging between 41 and 69 and signed in informed consent to participate in this trial voluntarily.
  The patients who do not use opioid medications immediately before the day of surgery for four weeks.

INTERVENTIONS:
Other: History for opioid use
  Arms: Chronic Opioid User

SUMMARY:
The purpose of this study is to find difference in Minimum Alveolar Concentration(MAC) for maintaining Bispectral Index (BIS) below 50 between chronic opioid users and opioid naive patients.

DETAILED DESCRIPTION:
1. Patients selection in elective surgery which need general anesthesia.
2. MAC BIS50 data was collected in each patients (by blinded investigator)
3. The data collection will be continued for enough sample size for using Dixon Up Down Method Analysis
4. After Data collection, MAC BIS below 50 will be analyzed in both groups ( Chronic opioid users versus opioid naive patients)

ELIGIBILITY:
Inclusion Criteria:

* The patients(ASA class I-III) who receive elective surgery
* signed in informed consent to participate in this trial voluntarily.

Exclusion Criteria:

* History of Monoamine Oxidase (MAO) inhibitor use
* Chronic alcoholics
* Acute alcohol abuser
* Contraindication for inhalation agent use (Sevoflurane)
* BMI >30
* History of medication use, which affect in the minimum concentration of sevoflurane;(barbiturates, chlorpromazine, diazepam, hydroxyzine, verapamil, marijuana)
* Craniotomy

Ages: 41 Years to 69 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2015-06; Primary Completion 2015-12 (Estimated); Study Completion 2016-06 (Estimated)

PRIMARY OUTCOMES:
Minimum Alveolar Concentration below BIS 50 in Sevoflurane; percentage (eg: 1.2%) | 15 minutes after pre-set of the concentration of sevoflurane
  Dixon's up down method is applied in this study. So pre-set concentration of sevoflurane will be used in each group.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anesthesiology and Pain Medicine, National Cancer Center, Goyang-si, Gyeonggi-do 10408, South Korea

REFERENCES:
- [Background] Matsuura T, Oda Y, Tanaka K, Mori T, Nishikawa K, Asada A. Advance of age decreases the minimum alveolar concentrations of isoflurane and sevoflurane for maintaining bispectral index below 50. Br J Anaesth. 2009 Mar;102(3):331-5. doi: 10.1093/bja/aen382. Epub 2009 Jan 24. PMID 19168857
- [Derived] Oh TK, Eom W, Yim J, Kim N, Kwon K, Kim SE, Kim DH. The Effect of Chronic Opioid Use on End-Tidal Concentration of Sevoflurane Necessary to Maintain a Bispectral Index Below 50: A Prospective, Single-Blind Study. Anesth Analg. 2017 Jul;125(1):156-161. doi: 10.1213/ANE.0000000000001791. PMID 28614132